CLINICAL TRIAL: NCT03250806
Title: Early Detection of Aortic Stenosis in the Community: Role of Clinical and Echocardiographic Screening During Influenza Vaccination Multi-center, Prospective, Observational Cohort Study
Brief Title: Early Detection of Aortic Stenosis in the Community During Flu Vaccination
Acronym: FluClinic
Status: Completed | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: FluClinic
Record Dates: First submitted 2017-03-01; First posted 2017-08-16 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Aortic Stenosis
Keywords: aortic stenosis, auscultation, target echocardiography
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- newly identified aortic stenosis: Patients identified on auscultation or target echocardiography with aortic stenosis. Consecutive patients per centre with no limit to numbers.

SUMMARY:
Prospective cohort study to test the hypothesis that patients identified with severe aortic stenosis are under-diagnosed and under-treated. Such patients shall be identified by auscultation or target echocardiography during flu vaccination. The hypothesis is that this will increase detection of aortic stenosis in the community.

DETAILED DESCRIPTION:
The design plans for two study phases:

1. Feasibility study: screening by auscultation and target echocardiography during flu vaccination in a single practice in Birmingham;
2. Screening study: multi-centre screening by auscultation or target echocardiography in geographically diverse general practices across the United Kingdom.

In each phase, the patient will be identified by auscultation and target echocardiography. Management and onward referral will be at the clinical discretion of the GP. Results of clinical review, investigation, follow-up and management will be recorded at 3 months from that date.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged over 65years attending for influenza vaccination.
* written informed consent to data collection

Exclusion Criteria:

* known aortic stenosis
* previous aortic valve repair/replacement

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients identified on auscultation or target echocardiography with aortic stenosis. Consecutive patients per centre with no limit to numbers.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
prevalence of aortic stenosis | From date of examination until follow-up after three months
  Determination of the prevalence of aortic stenosis detected on screening performed during flu vaccination.
comparison of detection rate of aortic stenosis | From date of examination until follow-up after three months
  Comparison of detection rates of aortic stenosis using target auscultation vs detection by target 2D echocardiography.

SECONDARY OUTCOMES:
Evaluation of qualitative estimation of calcium burden on 2D echocardiography as a marker of AS severity | three months
  Method evaluation
Calculation of costs in screening with auscultation versus target 2DE in screening for AS to inform future cost-efficacy studies of screening for AS. | three months
  Cost evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Richard Steeds, MD, Principal Investigator — Queen Elizabeth Hospital, Birmingham, UK; Peter Bramlage, MD, Study Chair — IPPMed UK Ltd
Locations (2):
- United Kingdom (2):
  - Whaddon Medical Center, Milton Keynes, Buckinghamshire
  - Swanswell Medical Centre, Birmingham

IPD SHARING:
Plan to Share IPD: No